CLINICAL TRIAL: NCT01032447
Title: Overcoming Obstacles to Clinical Trials Enrollment Through a Navigator Program
Status: Terminated | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Other Study IDs: GYN0001; GYN0001 (Other: Stanford University); SU-10262009-4240 (Other: Stanford)
Record Dates: First submitted 2009-12-11; First posted 2009-12-15 (Estimated); Last update posted 2016-09-28 (Estimated); Status verified 2016-09

CONDITIONS: Genital Neoplasms, Female; Gynecologic Cancers; Breast Cancer
MeSH Terms: conditions — Genital Neoplasms, Female; Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: Navigator Support — Standard of Care
  Other Names: ULACC Navigator Training Program

SUMMARY:
Pilot study for assessing the effectiveness of a Navigator program to aid in clinical trial participation amongst the Chinese demographic

ELIGIBILITY:
Inclusion Criteria:

Cancer patients for Focus Group must meet the following criterion:

* diagnosis of any gynecologic or breast cancer and be pursuing treatment here at Stanford within the last 2 years
* must read and speak Chinese
* willing and able to participant in group discussions

Cancer patients to receive Navigator Support must meet the following criterion:

* Newly diagnosed with gynecologic or breast cancer -pursuing treatment at Stanford Cancer Center
* must read and speak Chinese
* willing and able to have an individual relationship with a Navigator

Health Professional must meet the following criterion:

-must currently work in the Stanford gynecologic Oncology Clinic

Navigators must meet the following criterion:

* Chinese and English speaking
* willing and able to participate in training and to serve as a Navigator
* preferably a Cancer survivor

Exclusion Criteria:

Cancer patients must have a GOG performance status of 0-2 (see attached document for further details). Focus Group participate MAY be able to be participating in another study but patients who are already participating in a clinical trial will not be assigned a Navigator.

No Exclusionary criterion for Health Professionals or Navigators.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: diagnosis of any gynecologic or breast cancer and be pursuing treatment here at Stanford within the last 2 years
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2010-01; Primary Completion 2011-01 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
feasibility of the program | one year

CONTACTS AND LOCATIONS:
Overall Officials: Nelson N Teng, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States